CLINICAL TRIAL: NCT06621472
Title: Retrolaminar Block Versus Subcostal Transversus Abdominis Plane Block in Patients Undergoing Open Liver Resection Surgery
Brief Title: Retrolaminar Block Versus Subcostal Transversus Abdominis Plane Block in Liver Resection Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sayed Mahmoud Abed, assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: analgesia in hepatectomy
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Cancer Liver
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Tea

STUDY DESIGN:
Intervention Model Description: double blind
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- • Group R: Retrolaminar block (RLB) (Experimental): Patients will receive bilateral ultrasound guided retrolaminar block with injection of 20 ml bupivacaine 0.25% in each side.
  Interventions: Procedure: Retrolaminar block group
- Group T. Subcostal transversus abdominis plane block (STAP) (Experimental): Patients will receive bilateral Ultrasound guided subcostal TAP with injection of 20 ml bupivacaine 0.25% in each side.
  Interventions: Other: subcostal TAP technique
- Epidural (Experimental): By loss of resistant technique and catheter insertion at the level of thoracic vertebrae (7-10)
  Interventions: Other: thoracic Epidural

INTERVENTIONS:
Procedure: Retrolaminar block group — patients will be placed in a sitting position. The transducer will be positioned vertically 3 cm lateral to the midline at the level of the 7th thoracic transverse process. The muscles of the back, the transverse process, and the pleura between two transverse processes will be visualized. The needle will be introduced in a cranial-caudal direction toward the lamina using the in-plane method until the tip lay in the lamina 1 mL of normal saline will be injected to confirm the correct needle tip position by visualizing the spread. After negative aspiration, 20 mL of 0.25% isobaric bupivacaine. The procedure will be repeated on the opposite side.
  Arms: • Group R: Retrolaminar block (RLB)
Other: subcostal TAP technique — The transducer will be placed obliquely along the subcostal margin near the xiphisternum in the midline of the abdomen. The rectus abdominis muscle and underlying transversus abdominis muscle will be identified. The position of the transversus abdominis muscle will be confirmed by sliding the transducer laterally until the aponeuroses of the external and internal oblique muscle will be visualized. The transversus abdominis muscle will be then identified, being posterior to the internal oblique muscle and will be followed back medially to confirm its position beneath the rectus muscle. the needle will be introduced through the rectus muscle in a superomedial-to-inferolateral direction towards the transversus abdominis muscle using the in-plane method, and 20 mL of 0.25% isobaric bupivacaine will be injected
  Arms: Group T. Subcostal transversus abdominis plane block (STAP)
Other: thoracic Epidural — Before induction of general anesthesia the epidural catheter was inserted under sterile condition with a loss of resistance technique by an 18G needle at a mid-thoracic level (Th 7-10) to cover the dermatomes innervating the incision in the upper abdomen. The epidural infusion consisting of bupivacaine 1 mg/mL, and fentanyl 2 μg/mL was activated on the attending anesthesiologist's decision. Following the hospital protocols, the infusion rate was initiated at 5-10 mL/h, increased to maximum 15 mL/h if necessary, bolus dose of 5 mL was allowed every 30 minutes.
  Arms: Epidural

SUMMARY:
Adequate pain control improves postoperative outcomes and is imperative for enhanced recovery after surgery (ERAS) . Open liver resection surgery is associated with intraoperative blood loss, hypotension, coagulopathy, pulmonary complications, liver impairment, and renal impairment, making perioperative pain management challenging . Multimodal analgesic strategies employing regional techniques decrease postoperative pain and opioid consumption following liver resections. Thoracic epidural analgesia (TEA) is considered the 'gold standard' for open thoracic and abdominal surgical procedures .

DETAILED DESCRIPTION:
The retrolaminar block (RLB) is a modified paravertebral block that administers local anesthetic between the lamina of the thoracic vertebra and the erector spinae muscles, using landmark technique or under ultrasound guidance, rather than entering the needle into the thoracic paravertebral space (TPVS) directly. Moreover, real-time ultrasound guidance can help identify the lamina and monitor the spread of local anesthetic .

Ultrasound-guided Subcostal Transversus Abdominis Plane (TAP) Block is proven to provide adequate analgesia for upper and lower abdominal surgeries. A local anesthetic (LA) is deposited in the plane between the transversus abdominis and posterior sheath of the rectus muscle in the subcostal region to anesthetize the anterior cutaneous branches of the lower intercostal nerves (T7-T11). In this study, we aimed to compare the analgesic effect of RLB and subcostal TAP block in patients undergoing open liver resection surgery.

ELIGIBILITY:
Inclusion Criteria:

Physical status American Society of Anesthesiologists (ASA)II, III. Body mass index (BMI): 20-35 kg/m2.

Exclusion Criteria:

Patient refusal Physical status ASA IV BMI < 20 kg/m2 and >35 kg/m2 known sensitivity or contraindication to drug used in the study (local anesthetics, opioids).

History of psychological disorders and/or chronic pain. Contraindication to regional anesthesia e.g., local sepsis, pre- existing peripheral neuropathies, and coagulopathy.

Severe respiratory, cardiac disorders and renal disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
post-operative analgesic consumption for 24 hours among study groups. | for 24 hours postoperative
  measuring total dose of narcotics required for the patient in study groups

CONTACTS AND LOCATIONS:
Overall Officials: sayed M Abed, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
shared through web
Supporting Information: Study Protocol
Time Frame: starting in march 2025
Access Criteria: web

REFERENCES:
- [Background] Joshi GP, Kehlet H. Postoperative pain management in the era of ERAS: An overview. Best Pract Res Clin Anaesthesiol. 2019 Sep;33(3):259-267. doi: 10.1016/j.bpa.2019.07.016. Epub 2019 Jul 25. PMID 31785712
- See also: Agarwal V, Divatia JV: Enhanced recovery after surgery in liver resection: current concepts and controversies. Korean J Anesthesiol. 2019, 72:119-29. 10.4097/kja.d.19.00010 — https://pubmed.ncbi.nlm.nih.gov/30841029/